CLINICAL TRIAL: NCT04694573
Title: Collaborative Transplant Study (CTS) Pre- and Post-Transplantation Covid-19 Serum Studies: Antibody Development Following a SARS-CoV-2 Infection
Brief Title: Multicenter CTS Pre-and Post-Transplantation Covid-19 Serum Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Caner Suesal, Professor, Institute of Immunology, Heidelberg University
Other Study IDs: CTS Covid-19 Serum Studies
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Kidney Transplant; Complications; Kidney Transplant Failure and Rejection; Liver Transplant; Complications; Liver Transplant Failure and Rejection
Keywords: Covid-19; SARS-CoV-2; Kidney Transplantation; Liver Transplantation; donor-specific antibodies; dnDSA
MeSH Terms: conditions — COVID-19; Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Serum; EDTA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- POST-TX Covid-19 Serum Study Case: Kidney or liver-transplanted patients being hospitalized due to an infection with SARS-CoV-2
- POST-TX Covid-19 Serum Study Control: 2 matched controls without SARS-CoV-2 infection after TX; matching according to
  * age (18-34, 35-59, 60-75 years)
  * sex
  * type of transplantation
  * time after transplantation (0-180, 181-365, 366-1095, 1096-2555, >2555 days after TX)
- PRE-TX Covid-19 Serum Study Case: Patients being kidney or liver-transplanted after having had an infection with SARS-CoV-2
- PRE-TX Covid-19 Serum Study Control: 2 matched controls without SARS-CoV-2 infection prior to TX; matching according to
  * age(18-34, 35-59, 60-75 years)
  * sex
  * type of transplantation

SUMMARY:
The Covid-19 Serum Study is a prospective case-control study in

1. kidney or liver transplanted patients being hospitalized due to an infection with Severe Acute Respiratory Syndrome Coronavirus Type 2 (SARS-CoV-2) after transplantation (TX) (POST-TX Covid-19 Serum Study)

   or
2. patients receiving kidney or liver transplantation after having had a SARS-CoV-2 infection (PRE-TX Covid-19 Serum Study)

The aim of this study is to evaluate the development of de novo donor specific antibodies (dnDSA) in transplanted patients being hospitalized due to an infection with SARS-CoV-2 (POST-TX Covid-19 Serum Study) as well as in patients receiving kidney or liver transplantation after having had an infection with SARS-CoV-2 prior to transplantation (PRE-TX Covid-19 Serum Study).

Further, the investigators will evaluate possible consequences of having had a SARS-CoV-2 infection prior or after liver or kidney transplantation with regard to graft survival and incidence of graft rejection episodes as well as SARS-CoV-2 specific antibody development after SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Kidney-transplant recipients and full-size liver-recipients (de-novo or re-transplanted)
* Participant or legal guardian is willing and able to give informed consent for participation in the trial
* SARS-CoV-2 infection before transplantation (PRE-TX Covid-19 Serum Study) or after transplantation (POST-TX Covid-19 Serum Study)

Specific Inclusion Criteria for PRE-TX Covid-19 Serum Study:

* Kidney or liver transplantation between Dec 17,2020 - Dec 17, 2021

Specific Inclusion Criteria for POST-TX Covid-19 Serum Study:

* Hospitalization due to SARS-CoV-2 infection in between Dec 17,2020 - Dec 17, 2021

Exclusion Criteria:

* Participants not meeting the inclusion criteria
* multi-organ transplant recipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney- or liver transplant recipients with a SARS-CoV-2 infection prior to transplantation (PRE-TX Covid-19 Serum Study) or a SARS-CoV-2 infection after transplantation (POST-TX Covid-19 Serum Study), 2 matched controls
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in dnDSA development (PRE-TX Covid-19 Serum Study) | Year 1, 2, 3, 5 after day of transplantation
Change in dnDSA development (POST-TX Covid-19 Serum Study) | at day 60-90 after being hospitalized due to Covid-19; 1,2,3,5 years after day of hospitalization due to Covid-19
Graft Survival (PRE-TX Covid-19 Serum-Study) | Year 1, 2, 3, 5 after day of transplantation
Graft Survival (Post-TX Covid-19 Serum-Study) | at day 60-90 after being hospitalized due to Covid-19; 1,2,3,5 years after day of hospitalization due to Covid-19

SECONDARY OUTCOMES:
Incidence of graft rejection (PRE-TX Covid-19 Serum Study) | Year 1, 2, 3, 5 after day of transplantation
Incidence of graft rejection (POST-TX Covid-19 Serum Study) | at day 60-90 after being hospitalized due to Covid-19; 1,2,3,5 years after day of hospitalization due to Covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Caner Suesal, Professor, Principal Investigator — Institute of Immunology Heidelberg; Christian Morath, Professor, Principal Investigator — Department of Nephrology, Heidelberg
Locations (1):
- Nierenzentrum Heidelberg, Heidelberg, DE, Germany